CLINICAL TRIAL: NCT07065383
Title: Intramyocellular Lipid Compartments After Glucagon-like Peptide 1 Receptor Agonist Therapy in Type 2 Diabetes - Rebalancing the Fat Content of the Heart and Muscles
Brief Title: Rebalancing the Fat Content of the Heart and Muscles
Acronym: Re-CHARM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Grampian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 3-034-24
Record Dates: First submitted 2025-06-24; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — semaglutide; Endurance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Semaglutide administration plus dietary counselling and physical activity encouragement (Placebo Comparator): Semaglutide administration plus dietary counselling and physical activity encouragement
  Interventions: Drug: Semaglutide administration plus dietary counselling and physical activity encouragement
- Semaglutide and supervised training program (Active Comparator): Semaglutide administration plus a personalised and supervised program of resistance and endurance training
  Interventions: Drug: Semaglutide plus a personalised and supervised program of resistance and endurance training

INTERVENTIONS:
Drug: Semaglutide administration plus dietary counselling and physical activity encouragement — Semaglutide administration plus dietary counselling and physical activity encouragement
  Other Names: Semaglutide with dietary counselling and physical activity encouragement
  Arms: Semaglutide administration plus dietary counselling and physical activity encouragement
Drug: Semaglutide plus a personalised and supervised program of resistance and endurance training — Semaglutide administration plus a personalised and supervised program of resistance and endurance training.
  Other Names: Semaglutide plus personalised and supervised resistance and endurance training program
  Arms: Semaglutide and supervised training program

SUMMARY:
Traditional diabetes therapies focus on improving blood sugar control. However, many studies show that this may not be enough. New treatments focusing on weight loss have heralded better results. One of these treatments is Semaglutide and the investigators wish to examine its effects further in this study. The investigators propose to investigate what happens to the fat inside the heart and the leg muscles.

DETAILED DESCRIPTION:
Traditionally, diabetes therapies focus on improving glycaemic control. However, decades of well conducted clinical trials showed that glycaemic control alone has failed to reduce both all-cause and cardiovascular mortality in diabetes patients. The new diabetes treatment strategies of combining glucose control with weight reduction have heralded better cardiovascular outcomes, however their follow-up has been relatively short-term.

The investigators propose to explore the effects of semaglutide administration plus dietary counselling and physical activity encouragement versus a more intensive strategy of semaglutide administration plus a personalised and supervised program of resistance and endurance exercise training.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a confirmed diagnosis of type 2 diabetes established in the previous 10 years between the ages of 20 and 75
* HbA1c ≥ 53 mmol/mol (7%) typically on diet and/or metformin/sulphonylureas (and/or sodium-glucose cotransporter-2 inhibitors, Dipeptidyl peptidase 4 inhibitors, thiazolidinediones, but not on insulin)
* Patients who do not meet the WHO recommendations on physical activity (≤150 minutes per week) of moderate-vigorous physical activity (MVPA)
* Patients who have a BMI of ≥27 but with a body weight of less than 140kgs due to limitations of the scanner table weight limit
* Current or recent (within 3 months) eGFR >30 mL/min/1.73m2)
* Able to understand written and spoken English

Exclusion Criteria:

* Any previously unknown cardiac condition other than mild valvular disease
* Any history of known coronary artery disease (including myocardial infarction and myocardial infarction with normal coronary arteries)
* Any relevant or untreated endocrine condition (i.e. Cushings)
* Impaired renal function (defined as estimated glomerular filtration rate of less than 30 mL/min/1.73m2)
* Blood pressure of more than 180/100 mmHg
* Patients on any other medication known to influence glucose or fatty acids metabolism (niacin, omega-3 fatty acids, other glucagon-like peptide-1 receptor agonists)
* Patients with any dietary habits that may interfere with the investigation (for example high fat vegan diets, as we know form prior research that they have very different intramyocellular fat storage compared to those on no dietary preferences)
* Patients with any history of any medical or surgical condition that in the judgement of the investigators may interfere with the exercise regime (i.e. peripheral vascular disease, arthritis), fatty acids metabolism (i.e. lipid storage diseases) or may compromise the safety of the participant (i.e. neurological syndromes for whom an intense exercise program could result in musculo-skeletal injury or accidents due to loss of balance).
* Patients with a sensitivity to Semaglutide (known hypersensitivity, diabetic retinopathy, pregnancy, history of pancreatitis or history of any cancer)
* Significant asthma or pulmonary disease
* Participants unable to cycle on the ergometer
* Unable to perform exercise testing (e.g. prosthetic limbs)
* Pregnancy, breastfeeding or considering pregnancy.
* Patients who have recently had gastrointestinal contrast or radionuclides
* Inability to lie flat or remain motionless for scanning procedures
* Patients whose girth size cannot allow them to fit in the magnetic resonance scanner (there is no set location to measure as this is different for everyone, but we have a plastic hoop that can be fitted around the largest circumference to check the fit)
* Subjects who are not able to engage into a physical training regime or feel that they do not have the interest or sustained motivation to follow one.
* Participants currently enrolled in other interventional clinical research
* Participants not able to understand written or verbal English

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
1H-magnetic resonance spectroscopy | From enrollment to the end of treatment at the end of 12 weeks
  Non-invasive proton magnetic resonance spectroscopy (1H MRS) for assessment to determine the total intramyocellular fat

SECONDARY OUTCOMES:
Intramyocellular lipid pool compartments | From enrollment to the end of treatment at the end of 12 weeks
  Intramyocellular Lipid pool compartments examined with non-invasive proton magnetic resonance spectroscopy (1H MRS) and turnover examined with stable isotopes

CONTACTS AND LOCATIONS:
Overall Officials: Dana Dawson, DM, Principal Investigator — University of Aberdeen

IPD SHARING:
Plan to Share IPD: No
Anonymised data will be made available through request at time of publication depending on journal requirements.

REFERENCES:
- [Background] Rodriguez-Gutierrez R, Montori VM. Glycemic Control for Patients With Type 2 Diabetes Mellitus: Our Evolving Faith in the Face of Evidence. Circ Cardiovasc Qual Outcomes. 2016 Sep;9(5):504-12. doi: 10.1161/CIRCOUTCOMES.116.002901. Epub 2016 Aug 23. PMID 27553599
- [Background] von Gerichten J, West AL, Irvine NA, Miles EA, Calder PC, Lillycrop KA, Fielding BA, Burdge GC. The Partitioning of Newly Assimilated Linoleic and alpha-Linolenic Acids Between Synthesis of Longer-Chain Polyunsaturated Fatty Acids and Hydroxyoctadecaenoic Acids Is a Putative Branch Point in T-Cell Essential Fatty Acid Metabolism. Front Immunol. 2021 Oct 5;12:740749. doi: 10.3389/fimmu.2021.740749. eCollection 2021. PMID 34675928
- [Background] Burdge GC, Wright P, Jones AE, Wootton SA. A method for separation of phosphatidylcholine, triacylglycerol, non-esterified fatty acids and cholesterol esters from plasma by solid-phase extraction. Br J Nutr. 2000 Nov;84(5):781-7. PMID 11177194
- [Background] FOLCH J, LEES M, SLOANE STANLEY GH. A simple method for the isolation and purification of total lipides from animal tissues. J Biol Chem. 1957 May;226(1):497-509. No abstract available. PMID 13428781
- [Background] Johnson NA, Walton DW, Sachinwalla T, Thompson CH, Smith K, Ruell PA, Stannard SR, George J. Noninvasive assessment of hepatic lipid composition: Advancing understanding and management of fatty liver disorders. Hepatology. 2008 May;47(5):1513-23. doi: 10.1002/hep.22220. PMID 18393289
- [Background] Boesch C, Slotboom J, Hoppeler H, Kreis R. In vivo determination of intra-myocellular lipids in human muscle by means of localized 1H-MR-spectroscopy. Magn Reson Med. 1997 Apr;37(4):484-93. doi: 10.1002/mrm.1910370403. PMID 9094069
- [Background] Scally C, Abbas H, Ahearn T, Srinivasan J, Mezincescu A, Rudd A, Spath N, Yucel-Finn A, Yuecel R, Oldroyd K, Dospinescu C, Horgan G, Broadhurst P, Henning A, Newby DE, Semple S, Wilson HM, Dawson DK. Myocardial and Systemic Inflammation in Acute Stress-Induced (Takotsubo) Cardiomyopathy. Circulation. 2019 Mar 26;139(13):1581-1592. doi: 10.1161/CIRCULATIONAHA.118.037975. PMID 30586731
- [Background] Wallace TM, Levy JC, Matthews DR. Use and abuse of HOMA modeling. Diabetes Care. 2004 Jun;27(6):1487-95. doi: 10.2337/diacare.27.6.1487. PMID 15161807
- [Background] Fillmer A, Hock A, Cameron D, Henning A. Non-Water-Suppressed 1H MR Spectroscopy with Orientational Prior Knowledge Shows Potential for Separating Intra- and Extramyocellular Lipid Signals in Human Myocardium. Sci Rep. 2017 Dec 4;7(1):16898. doi: 10.1038/s41598-017-16318-0. PMID 29203776
- [Background] Blundell J, Finlayson G, Axelsen M, Flint A, Gibbons C, Kvist T, Hjerpsted JB. Effects of once-weekly semaglutide on appetite, energy intake, control of eating, food preference and body weight in subjects with obesity. Diabetes Obes Metab. 2017 Sep;19(9):1242-1251. doi: 10.1111/dom.12932. Epub 2017 May 5. PMID 28266779
- [Background] Wilding JPH, Batterham RL, Calanna S, Davies M, Van Gaal LF, Lingvay I, McGowan BM, Rosenstock J, Tran MTD, Wadden TA, Wharton S, Yokote K, Zeuthen N, Kushner RF; STEP 1 Study Group. Once-Weekly Semaglutide in Adults with Overweight or Obesity. N Engl J Med. 2021 Mar 18;384(11):989-1002. doi: 10.1056/NEJMoa2032183. Epub 2021 Feb 10. PMID 33567185
- [Background] Lincoff AM, Brown-Frandsen K, Colhoun HM, Deanfield J, Emerson SS, Esbjerg S, Hardt-Lindberg S, Hovingh GK, Kahn SE, Kushner RF, Lingvay I, Oral TK, Michelsen MM, Plutzky J, Tornoe CW, Ryan DH; SELECT Trial Investigators. Semaglutide and Cardiovascular Outcomes in Obesity without Diabetes. N Engl J Med. 2023 Dec 14;389(24):2221-2232. doi: 10.1056/NEJMoa2307563. Epub 2023 Nov 11. PMID 37952131
- [Background] Marso SP, Bain SC, Consoli A, Eliaschewitz FG, Jodar E, Leiter LA, Lingvay I, Rosenstock J, Seufert J, Warren ML, Woo V, Hansen O, Holst AG, Pettersson J, Vilsboll T; SUSTAIN-6 Investigators. Semaglutide and Cardiovascular Outcomes in Patients with Type 2 Diabetes. N Engl J Med. 2016 Nov 10;375(19):1834-1844. doi: 10.1056/NEJMoa1607141. Epub 2016 Sep 15. PMID 27633186
- [Background] Iacobellis G. Epicardial adipose tissue in contemporary cardiology. Nat Rev Cardiol. 2022 Sep;19(9):593-606. doi: 10.1038/s41569-022-00679-9. Epub 2022 Mar 16. PMID 35296869
- [Background] Dube JJ, Amati F, Stefanovic-Racic M, Toledo FG, Sauers SE, Goodpaster BH. Exercise-induced alterations in intramyocellular lipids and insulin resistance: the athlete's paradox revisited. Am J Physiol Endocrinol Metab. 2008 May;294(5):E882-8. doi: 10.1152/ajpendo.00769.2007. Epub 2008 Mar 4. PMID 18319352
- [Background] Goodpaster BH, He J, Watkins S, Kelley DE. Skeletal muscle lipid content and insulin resistance: evidence for a paradox in endurance-trained athletes. J Clin Endocrinol Metab. 2001 Dec;86(12):5755-61. doi: 10.1210/jcem.86.12.8075. PMID 11739435
- [Background] Bergman BC, Perreault L, Hunerdosse DM, Koehler MC, Samek AM, Eckel RH. Increased intramuscular lipid synthesis and low saturation relate to insulin sensitivity in endurance-trained athletes. J Appl Physiol (1985). 2010 May;108(5):1134-41. doi: 10.1152/japplphysiol.00684.2009. Epub 2010 Mar 18. PMID 20299618
- [Background] Petersen KF, Dufour S, Morino K, Yoo PS, Cline GW, Shulman GI. Reversal of muscle insulin resistance by weight reduction in young, lean, insulin-resistant offspring of parents with type 2 diabetes. Proc Natl Acad Sci U S A. 2012 May 22;109(21):8236-40. doi: 10.1073/pnas.1205675109. Epub 2012 Apr 30. PMID 22547801
- [Background] Amati F, Dube JJ, Alvarez-Carnero E, Edreira MM, Chomentowski P, Coen PM, Switzer GE, Bickel PE, Stefanovic-Racic M, Toledo FG, Goodpaster BH. Skeletal muscle triglycerides, diacylglycerols, and ceramides in insulin resistance: another paradox in endurance-trained athletes? Diabetes. 2011 Oct;60(10):2588-97. doi: 10.2337/db10-1221. Epub 2011 Aug 26. PMID 21873552
- [Background] Levelt E, Mahmod M, Piechnik SK, Ariga R, Francis JM, Rodgers CT, Clarke WT, Sabharwal N, Schneider JE, Karamitsos TD, Clarke K, Rider OJ, Neubauer S. Relationship Between Left Ventricular Structural and Metabolic Remodeling in Type 2 Diabetes. Diabetes. 2016 Jan;65(1):44-52. doi: 10.2337/db15-0627. Epub 2015 Oct 5. PMID 26438611
- [Background] Ozasa N, Furukawa Y, Morimoto T, Tadamura E, Kita T, Kimura T. Relation among left ventricular mass, insulin resistance, and hemodynamic parameters in type 2 diabetes. Hypertens Res. 2008 Mar;31(3):425-32. doi: 10.1291/hypres.31.425. PMID 18497461
- [Background] Summers SA, Nelson DH. A role for sphingolipids in producing the common features of type 2 diabetes, metabolic syndrome X, and Cushing's syndrome. Diabetes. 2005 Mar;54(3):591-602. doi: 10.2337/diabetes.54.3.591. PMID 15734832
- [Background] Dube JJ, Amati F, Toledo FG, Stefanovic-Racic M, Rossi A, Coen P, Goodpaster BH. Effects of weight loss and exercise on insulin resistance, and intramyocellular triacylglycerol, diacylglycerol and ceramide. Diabetologia. 2011 May;54(5):1147-56. doi: 10.1007/s00125-011-2065-0. Epub 2011 Feb 17. PMID 21327867
- [Background] King DS, Dalsky GP, Clutter WE, Young DA, Staten MA, Cryer PE, Holloszy JO. Effects of exercise and lack of exercise on insulin sensitivity and responsiveness. J Appl Physiol (1985). 1988 May;64(5):1942-6. doi: 10.1152/jappl.1988.64.5.1942. PMID 3292505
- [Background] Cheng YJ, Imperatore G, Geiss LS, Saydah SH, Albright AL, Ali MK, Gregg EW. Trends and Disparities in Cardiovascular Mortality Among U.S. Adults With and Without Self-Reported Diabetes, 1988-2015. Diabetes Care. 2018 Nov;41(11):2306-2315. doi: 10.2337/dc18-0831. Epub 2018 Aug 21. PMID 30131397